CLINICAL TRIAL: NCT03051321
Title: Maintaining Lower Levels of Care Through Automated Perineal Hygiene
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: SchwabCare (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SC-02
Record Dates: First submitted 2017-02-07; First posted 2017-02-13 (Actual); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Incontinence; Dermatitis
MeSH Terms: conditions — Dermatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Wellness toileting system (Experimental): Subjects given SchwabCare Wellness Toileting system
  Interventions: Device: Wellness toilet system

INTERVENTIONS:
Device: Wellness toilet system — Water-based toileting with capacity to apply zinc oxide barrier spray to treat incontinence associated dermatitis
  Other Names: SchwabCare Wellness Toileting System

SUMMARY:
The inability to independently manage perineal hygiene after toileting is a common issue for those in assisted living and nursing home environments. It is associated with skin breakdown (dermatitis), increased nursing costs, and loss of patient self-esteem and independence. Water-based toileting has been evaluated as a possible adjunct to patient care, but its uptake has been limited by ineffective cleansing and drying.

40 subjects with limitations in independent capacity for perineal hygiene that require assistance with toileting will be recruited from a continued care retirement center. Subjects will be assessed for incontinence, and skin breakdown or irritation. Subjects will be provided a Wellness Toilet System, cleanser, and, if needed, zinc oxide barrier spray to be applied in cases of dermatitis.

Investigators hypothesize that subjects given the device will remain more independent, with higher quality of life. Secondary hypotheses are that subjects will experience improved relationships with their caregivers, and that active dermatitis will be treated in those already with the condition, and prevented in those at risk.

DETAILED DESCRIPTION:
The prevalence of incontinence and inability to maintain personal perineal hygiene increases with higher levels of nursing care. While more than 75% of those in assisted living and home care settings are able to independently care for themselves after toileting, up to 75% of nursing home residents have regular episodes of urinary or fecal incontinence and require aid with toileting. This implies that whereas incontinence is a primary diagnosis in only 10% of nursing home admissions, it represents a major contributor to morbidity among all nursing home residents, and with that, an important target for efforts at cost containment. Inadequate independent perineal hygiene and dependence on caregivers for effective toileting raises global costs and adversely affects well-being for those in assisted living and dependent living environments. It is also associated with an increase in incontinence and incontinence associated dermatitis, which carries higher risks of urinary tract infection and skin infection. Finally, in many institutions, loss of toileting independence mandates a shift to a higher intensity environment, and with that incurs significant cost.

Water-based toileting has been evaluated as a potential intervention for nursing home residents with impaired toileting capacity. In that study, while investigators found significant overall improvement those using the device, less than half were neither effectively cleaned nor dry at the end of use. Because of this limited reliability, currently available devices are not thought to offer enough significant advantages for routine use in nursing home settings.

Incontinence and incontinence associated dermatitis (IAD) is common among residents with impaired perineal hygiene and toileting. Adherence to prescribed medications and therapies directed at the perineum is a major barrier to regular use among those with fecal or urinary incontinence. Difficulty in accessing the perineum make adherence challenging to those with both full and limited mobility, often requiring assistance from a caregiver. The associated loss of independence and dignity are major detriments to quality of life. Novel formulations of zinc oxide, using aerosol based spray application, facilitate use and improve patient acceptance. In a 2014 nursing home based industry study, spray based zinc oxide was preferred by 80% of patients and caregivers, and improved treatment and prevention of IAD in 70% of the study participants.

Adequate cleansing and drying prior to the application of barrier products is key to effective prevention of skin breakdown. Water-based cleaning of the perineum after toileting has been demonstrated to improve hygiene over standard mechanical, paper-based cleansing, especially in those with limited mobility or incontinence. Evidence further demonstrates that the addition of pH balanced cleansers, applied without mechanical abrasion from cloths or wipes, advances hygiene and minimizes risk of secondary infection.

Study Aims

The aims of this study are to evaluate whether an automated delivery system for cleansing the perineum can keep subjects who would normally move to higher levels of assistance at lower levels of nursing care. A secondary aim will be to evaluate whether an automated hands-free application of zinc oxide barrier spray effectively treats and prevents incontinence associated dermatitis in a population with active or recurrent IAD. Finally, the study aims to demonstrate cost savings through a cost effectiveness analysis.

ELIGIBILITY:
Inclusion Criteria:

- Limitation of Activity of Daily Living - Toileting, requiring assistance, beginning stages of unmanaged incontinence. For the purposes of this study, toileting refers to maintenance of hygiene and ability to clean the perineum after urination or defecation. It does not include inability to transfer to a commode only.

Exclusion Criteria:

* Inability to obtain consent
* Weight over 300 pounds
* Prior pelvic radiation
* Pelvic Floor surgery within the 6 weeks prior to enrollment
* Active perineal infection
* Active chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-06 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Days Remaining in independent living environment | 24 weeks
  Subject does not require assistance for perineal hygiene that requires change of living environment

SECONDARY OUTCOMES:
Improved quality of life | 24 weeks
  Subject using device will experience improved quality of life derived from the quality of life in incontinence scale
Treatment and prevention of incontinence associated dermatitis | 24 weeks
  Device will treat existing, and prevent dermatitis in subjects with incontinence, evaluated using the Kennedy Scale

CONTACTS AND LOCATIONS:
Overall Officials: Richard S Tilson, MD MPH, Principal Investigator — Director of Clinical Investigation
Locations (2):
- United States (2):
  - The Canterbury, Rancho Palos Verdes, California
  - The Village at Marymount, Garfield Heights, Ohio

IPD SHARING:
Plan to Share IPD: No